CLINICAL TRIAL: NCT04798807
Title: Screening Nutritional Status of Hospitalized Patients With Nutritional Risk Screening 2002 and Subjective Global Assessment Tools
Brief Title: Screening Nutritional Status of Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Neşe Kaya, Investigator, TC Erciyes University
Other Study IDs: 2016/144
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Malnourishment
Keywords: Nutritional assessment; Nutritional Risk Screening 2002; Subjective Global Assessment.
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized non-critical services patients: Patients, who were hospitalized in the clinics (hematology, neurology, gastroenterology, nephrology, endocrine, pulmonary disease and cardiology) of Malatya Training and Research Hospital, were screened both Nutritional Risk Screening 2002 (NRS-2002) and Subjective Global Assessment (SGA) tools within the first days of admission to the patients.
  The nutritional status of patients categorized according the screening tools.
  Nutritional Risk Screening 2002 (NRS-2002) : The patients were classified as being nutritionally risk (NRS+): total score ≥ 3 or nutritionally risk-free (NRS-): total score < 3 according to NRS 2002 results.
  Subjective Global Assessment (SGA) The SGA screening provides three alternative categories for nutritional classification: well nourished (A); mild-to-moderately malnourished (B); or severely malnourished (C).
  Interventions: Diagnostic Test: Nutritional screening

INTERVENTIONS:
Diagnostic Test: Nutritional screening

SUMMARY:
This study investigated the results of the nutritional status of hospitalized patients with Nutritional Risk Screening 2002 (NRS-2002) and Subjective Global Assessment (SGA) screening and compared the effects of two screening method in predicting malnutrition.

DETAILED DESCRIPTION:
In the cross-sectional study demographic data, body mass index (BMI), length of hospital stay (LOS), and cause of hospitalization of hospitalized patients were recorded. For the nutritional assessment all patients were screened with NRS 2002 and SGA within the first days of admission to the patients. The primary predictors of interest in our study were the NRS 2002 and SGA results of patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* non-bed-dependent
* non-critİcal service patients

Exclusion Criteria:

* < 18 years old,
* hospitalized due to surgical operation,
* pregnant women,
* breastfeeding women,
* bed-dependent,
* suffered an advanced disease that required palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized in the clinics (hematology, neurology, gastroenterology, nephrology, endocrine, pulmonary disease and cardiology) of Malatya Training and Research Hospital between January 1 and August 30, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Identifying malnourishment according to the Nutritional Risk Screening 2002 | First 48 hours of hospitalization
  The results of the Nutritional Risk Screening 2002 (NRS-2002): The patients were classified as being nutritionally risk (NRS+): total score ≥ 3 or nutritionally risk-free (NRS-): total score < 3 according to NRS 2002 results.
Identifying malnourishment according to the Subjective Global Assessment (SGA) | First 48 hours of hospitalization
  The results of the Subjective Global Assessment (SGA): The SGA screening provides three alternative categories for nutritional classification: well nourished (A); mild-to-moderately malnourished (B); or severely malnourished (C).
Compare the results of two screening tools. | Through study completion, an average of 1 year
  Compare the results of NRS-2002 and SGA tools on predicting malnutrition and nutritional status of patients.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04798807/Prot_SAP_000.pdf